CLINICAL TRIAL: NCT00184067
Title: A Randomized Phase II Continuation Booster Trial After a Vaccine Combining Tyrosinase/GP100/MART-1 Peptides Emulsified With Montanide ISA 51 With or Without GM-CSF for Patients With Resected Stages IIB/C, III, and IV Melanoma
Brief Title: Continuation Booster Trial After a Vaccine Combining Tyrosinase/GP100/MART-1 Peptides Emulsified With Montanide ISA 51 With or Without GM-CSF for Patients With Melanoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Primary PI left institution
Sponsor: University of Southern California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 10M-03-8
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-01

CONDITIONS: Melanoma
MeSH Terms: conditions — Melanoma | interventions — montanide ISA 51

ARMS (2):
- Peptide vaccine with Montanide ISA 51 + GM-CSF (Experimental): Peptide vaccine with Montanide ISA 51 GM-CSF
  Interventions: Biological: Montanide ISA 51
- Peptide vaccine with Montanide ISA 51 (Active Comparator): Peptide vaccine with Montanide ISA 51
  Interventions: Biological: Montanide ISA 51

INTERVENTIONS:
Biological: Montanide ISA 51

SUMMARY:
This is a study of a melanoma vaccine. Study participants will have melanoma that invaded deeply and spread to lymph nodes or another location. Although the participants' melanoma has been removed, there is a greater than 1 out of 2 chance it will return. There will be approximately 40 subjects in this study. The patients will have already taken part in a melanoma vaccine study, and in this current study, they will continue to receive booster injections of a similar vaccine given for two additional years.

This study will test an experimental vaccine. The vaccine contains peptides which are fragments of substances made by most melanomas. The substances are tyrosinase, gpl00 and melanoma antigen recognized by T cells (MART-1). The vaccine also includes an assistant called Montanide ISA 51. The assistant stimulates the immune system. This study will also test the effects of a second assistant granulocyte-macrophage colony-stimulating factor (GM-CSF). All participants will receive the vaccine and assistant Montanide ISA 51, but only half will receive the assistant GM-CSF. The patients have a one in two chance of receiving the assistant called GM-CSF. The main purpose of this study is to find out if the booster injections increase the body's immunity to melanoma and prevent its level of immunity from getting lower over time. The investigators also wish to know if the GM-CSF increases the body's immunity to melanoma when given with the melanoma vaccine.

The vaccine and assistant Montanide ISA 51 are not approved by the Food and Drug Administration (FDA). The assistant GM-CSF is approved by the FDA to increase infection-fighting white blood cells after chemotherapy. It is not approved by the FDA for treatment of melanoma. However, the FDA is permitting the vaccine and the assistants to be tested in this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have completed protocol 10M-01-1 or 10M-00-4 are eligible for this study provided that:

  1. They have received all injections with evidence of an immune response.
  2. They have not experienced recurrence of the melanoma.
  3. Not more than twelve months have elapsed since the final injection on either protocol.
  4. They experienced no grade 3 or 4 toxicity attributed to the prior vaccine regimen.
* Serum creatinine of 2.0 mg/dl or less, total bilirubin of 2.0 mg/dl or less and SGOT/SGPT of 2.5 X institutional norm or less.
* Total whte blood cell (WBC) of 3,000 or more with at least 1500 granulocytes, hemoglobin of 9.0 gm/dl or more, and platelet count of 100,000 per cu mm or more.
* ECOG performance status of 0 or 1.
* Patients will be eligible for this trial if they have failed alpha-interferon, if it is felt to be contraindicated due to a pre-existing medical or psychiatric condition or if they have refused treatment with it.
* Ability to read, understand and willingness to sign an institutional review board (IRB)-approved informed consent.
* Patients who have had another malignancy but with no evidence of disease for greater than 5 years from accrual to the current trial will be eligible if it is felt they are likely to be cured. Patients with squamous or basal carcinoma of the skin or carcinoma in situ of the cervix that have been treated with curative intent can be accrued to this trial 30 days after treatment.

Exclusion Criteria:

* Patients who have undergone any other systemic therapy for their melanoma, including radiation therapy since completion of 10M-01-1 or 10M-00-4.
* Have major systemic infections like pneumonia or sepsis, coagulation or bleeding disorders, or other major medical illnesses of the gastrointestinal, cardiovascular or respiratory systems.
* Require systemic, ocular or inhaled corticosteroids.
* Pregnant or lactating, since the risk of autoimmune reactivity to tyrosinase, MART-1 or gp100 is felt to present a risk to the fetus or a breast feeding infant. Effective birth control for men and women is required during and for four months after the study is finished.
* Known to be positive for hepatitis BsAg, hepatitis C antibody or HIV antibody. Since cells removed for ex vivo handling and tissue culture cannot be virus positive, and the effects of melanoma peptides might be detrimental to HIV positive patients, patients positive for the above viruses will not be treated in this trial.
* Have had a known allergic reaction to GM-CSF, Montanide ISA 51 (IFA) or any of the peptides included in this protocol.
* Have a prior history of uveitis or autoimmune inflammatory eye disease, immune hemolytic anemia or other active autoimmune disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-05; Primary Completion 2007-04 (Actual); Study Completion 2009-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Weber, Principal Investigator — University of Southern California
Locations (1):
- USC/Norris Comprehensive Cancer Center, Los Angeles, California, United States